CLINICAL TRIAL: NCT01271959
Title: A Multicenter, Post-Market Follow-up Study of ChemoFx® Chemoresponse Assay in Solid Tumors - ChemoFx® Registry Study
Brief Title: A Study of ChemoFx® Chemoresponse Assay in Solid Tumors - ChemoFx® Registry Study
Status: Terminated | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PT-207
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Solid Organ Tumors
Keywords: Ovarian; Fallopian Tube; Peritoneal; Uterine Neoplasms; Vulva; Endometrial; Cervical; Lung; Carcinoid; Sarcoma; Mesothelioma; Adenocarcinoma; Colorectal; Breast; Assay; Chemotherapy; Recurrent; Refractory; Persistent; Chemoresponse
MeSH Terms: conditions — Uterine Neoplasms; Carcinoid Tumor; Sarcoma; Mesothelioma; Adenocarcinoma; Recurrence

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA, RNA, and proteomic research will be conducted on excess tissue cells.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to collect information from patient's medical records that had a test called ChemoFx® ordered and to understand how doctors may have used the results of the ChemoFx® to treat patients with cancer.

DETAILED DESCRIPTION:
While studies support the clinical use of ChemoFx® in cancer patients, additional data are needed to further assess the utilization of this product in clinical practice. Such post-market data and information could be employed for product improvement as well as for the development of standards and regulations. This is a multicenter registry study of 3,000 patients with solid tumors. The study is not randomized, nor is it interventional in that the treating physician is free to choose how to employ ChemoFx® results in the clinical management of individual patients. Sites will be selected by Precision's clinical trials team based on past commercial usage of ChemoFx®.

Subjects who may be enrolled in this study are those who have been diagnosed with a solid tumor malignancy and for whom ChemoFx® has been ordered. ChemoFx® is ordered through the normal commercial process and is therefore billed to the patient's medical insurance.

All subjects will be appropriately consented before any study-specific data are collected. A limited dataset of patient demographics, oncology history, and therapeutic intervention will be collected in addition to ChemoFx® assay usage. Subjects will be treated based on the medical judgment of their treating physician(s). Patient survival data will be collected up to five years following the ChemoFx® commercial order. Additional disease progression data may be collected by Precision's CRAs at participating sites.

Optional Cell Research

Informed consent will be obtained to document subject's consent to use excess cells remaining in Precisions' commercial laboratory for additional research. This portion of the study may involve DNA, RNA, and proteomic research. To ensure the anonymity of each subject, any identifiers that would link the sample to the subject will be removed. The samples would then have gene expression profiling and or quantitative protein expression analysis performed. The goal of the research would be to identify a set of informative genes, intermediaries, and proteins and develop predictive algorithm(s) that seek to link the expression level of the gene, gene signature, intermediary, or protein to the clinical outcome of the patient. This portion of the study does not require any additional subject procedures. Neither physicians nor their patients will receive the results of the research performed. Results will not be placed in the subjects health care records and will not affect their medical care.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of solid tumor malignancy;
* Medically indicated to receive chemotherapy;
* Fresh tissue submitted from the solid tumor malignancy for testing with the ChemoFx® assay after August, 2006;
* Final ChemoFx® assay report is available;
* Subject must be at least 18 years of age;
* Subject must sign and date an IRB approved ICF.

Exclusion Criteria:

* Enrolled in PT-103, PT-106, PT-206, PT-301, or PT-304;
* Pregnant or lactating subjects;
* Subjects are not indicated to receive chemotherapy for their disease;
* Subjects with psychiatric or addictive disorders that would preclude obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with solid tumor malignancies
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine physicians' rate of compliance with ChemoFx assay results in the treatment of subjects with solid tumors. | Analysis of assay-directed compliance will be conducted immediately after information is collected.
To investigate the association between the results of Precision's ChemoFx assay results and overall survival in subjects with solid tumors. | From date of first dose of on-study chemotherapy to date of death or last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Williams, M.D., Principal Investigator — Precision Therapeutics, Inc.
Locations (25):
- United States (25):
  - Cardio-Thoracic Surgeons, P.C., Birmingham, Alabama
  - Hematology Oncology Associates, Oakland, California
  - Collaborative Research Group, Boynton Beach, Florida
  - Broward Oncology Associates, P.A., Fort Lauderdale, Florida
  - The Center For Gynecologic Oncology, Hollywood, Florida
  - GYN Oncology of Miami, Miami, Florida
  - Miami International Surgical Services, Miami, Florida
  - Orlando Cardiovascular Institute PA, Orlando, Florida
  - Edward H. Kaplan, M.D. & Associates, Skokie, Illinois
  - Iowa Clinic, Des Moines, Iowa
  - Central Baptist Hospital Clinical Research Center, Lexington, Kentucky
  - Oncology Associates of West Kentucky, Paducah, Kentucky
  - Grand Blanc Surgical Specialist, Grand Blanc, Michigan
  - Albany Thoracic & Esophageal Surgery, Albany, New York
  - North Shore Hematology Oncology, East Setauket, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - Center for Clinical Research and Technology University Hospitals of Cleveland, Cleveland, Ohio
  - The Regional Cancer Center, Erie, Pennsylvania
  - Barry S Siller MD, Houston, Texas
  - Colorectal Surgical Associates, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Cancer Care Northwest, Spokane, Washington
  - Heiskell, King, Burns & Tallman Surgical Associates, Inc., Morgantown, West Virginia